CLINICAL TRIAL: NCT02251145
Title: A Single Centre, Open-Label, Randomised, Parallel, Multiple Dose Comparison of the Effects of Tipranavir 500 mg and Ritonavir 100 mg or Tipranavir 750 mg and Ritonavir 200 mg Twice a Day for 11.5 Days on the Pharmacokinetic Characteristics of Tenofovir Disoproxil Fumarate 300 mg in Healthy Volunteers
Brief Title: Effects of Tipranavir (TPV) and Ritonavir (RTV) on the Pharmacokinetic Characteristics of Tenofovir Disoproxil Fumarate in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1182.46
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir; Tenofovir

ARMS (2):
- tipranavir/ritonavir low dose (Experimental)
  Interventions: Drug: Tipranavir low dose; Drug: Ritonavir low dose; Drug: Tenofovir disoproxil fumarate
- tipranavir/ritonavir high dose (Experimental)
  Interventions: Drug: Tipranavir high dose; Drug: Ritonavir high dose; Drug: Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Tipranavir low dose
  Arms: tipranavir/ritonavir low dose
Drug: Tipranavir high dose
  Arms: tipranavir/ritonavir high dose
Drug: Ritonavir low dose
  Arms: tipranavir/ritonavir low dose
Drug: Ritonavir high dose
  Arms: tipranavir/ritonavir high dose
Drug: Tenofovir disoproxil fumarate

SUMMARY:
Study to characterise the effects of two dose combinations of tipranavir/ritonavir (TPV 500 mg/RTV 100 mg and TPV 750 mg/RTV 200 mg) administered BID, on the pharmacokinetics of tenofovir disoproxil fumarate as well as the effects of tenofovir disoproxil fumarate on the pharmacokinetics of tipranavir/ritonavir.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to give written informed consent in accordance with institutional and regulatory guidelines and to comply with the investigational nature of the study and the related requirements
2. Healthy males or females between 18 and 60 years of age inclusive
3. A Body Mass Index >18.5 and <30 kg/m2
4. Ability to swallow numerous large capsules without difficulty
5. Reasonable probability for completion of the study, in the opinion of the investigator
6. Acceptable laboratory values that indicate adequate baseline organ function are required at the time of screening. Laboratory values are considered to be acceptable if severity <= Grade1 based on the AIDS Clinical Trials Group (ACTG) Division of AIDS (DAIDS) Grading Scale. All abnormal laboratory values > Grade 1 (e.g., creatine phosphokinase (CPK), amylase, triglycerides) are subject to approval by the BIPI clinical monitor. Cholesterol <= 240mg/dL at the time of screening is necessary for study entry
7. Acceptable medical history, physical examination and ECG are required prior to entering the study
8. Willingness to abstain from alcohol for 48 hours prior to Study Day 0 and abstain from alcohol for the duration of the study. In addition, Cabernet Sauvignon must not have been ingested within 15 days prior to Day 0 (Visit 2)
9. Willingness to abstain from ingesting grapefruit and grapefruit juice within 15 days of Day 0, Visit 2 and for the duration of the study
10. Willingness to abstain from ingesting Seville oranges, strawberries or strawberry extract, garlic supplements, St. John's Wort, Milk Thistle, or methylxanthine-containing drinks or food (coffee, tea, cola, energy drinks, chocolate, etc) within 72 hours of pharmacokinetic (PK) sampling days
11. Willingness to abstain from use of tobacco products for the duration of the study
12. Urine drug screen negative for illegal non-prescription drugs
13. Negative HIV serology
14. Negative for Hepatitis B surface antigen and Hepatitis C

Exclusion Criteria:

1. Female subjects who are of reproductive potential who:

   * Have a positive serum B-HCG at Visit 1 or 2 or
   * Have not been using regular oral contraception (combined oestrogen and progestogen pill or progestogen only pill) for 3 months and a barrier contraceptive method for at least 30 days prior to Visit 3 (Day 1) or a barrier contraceptive method for at least 3 months prior to Visit 3 (Day 1) or
   * Are not willing to use a reliable method of double-barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam)during the trial and 30 days after completion/termination or
   * Are breast-feeding
2. Participation in another trial with an investigational medicine for 30 days prior to Day 0 (Visit 2)
3. Ingestion of any known enzyme altering drug (such as phenothiazines, cimetidine, barbiturates, ketoconazole, fluconazole, rifampin, steroids, and herbal medications) for 30 days prior to Day 0 (Visit 2). Use of any other herbal/complementary treatment must be discussed in advance with the monitor and permission obtained prior to study entry
4. Ingestion of grapefruit, grapefruit juice, and Cabernet Sauvignon within 15 days prior to Day 0 (Visit 2)
5. Ingestion of Seville oranges, strawberries or strawberry extract, garlic supplements, St. John's Wort, Milk Thistle, or methylxanthine-containing drinks or food (coffee, tea, cola, energy drinks, chocolate, etc) within 72 hours of PK sampling days
6. Ingestion of antibiotics within 10 days prior to Day 0 (Visit 2)
7. Inability to comply with investigator's instructions
8. History of gastrointestinal, hepatic, or renal disorders within 60 days
9. History of alcohol abuse
10. Current use of cigarettes defined as greater than 10 cigarettes per day or rolling/pipe tobacco equivalent
11. Blood or plasma donations within 30 days prior to Day 0 (Visit 2)
12. Subjects with a seated systolic blood pressure either <100 mm Hg or >150 mm Hg; resting heart rate either <50 beats/min or >100 beats/min
13. Subjects with a history of any illness or allergy that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering tipranavir or ritonavir or tenofovir disoproxil fumarate to the subject
14. Subjects who have had an acute illness within 2 weeks prior to Day 0 (Visit 2)
15. Subjects who are currently taking any over-the-counter drug within 7 days prior to Day 0, (Visit 2) or who are currently taking any prescription drug that, in the opinion of the investigator in consultation with the clinical monitor and pharmacokineticist, might interfere with either the absorption, distribution or metabolism of the test substances
16. Hypersensitivity to tipranavir, ritonavir, or tenofovir disoproxil fumarate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2002-05; Primary Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration time curve from 0-24 hours (AUC0-24) for tenofovir | up to 24 hours
Area under plasma concentration time curve from 0-12hours (AUC0-12) for tipranavir/ritonavir | up to 12 hours
Maximum plasma concentration (Cmax) | up to 24 hours
Drug concentration in plasma at 12 hours after administration (C12h) for tenofovir | up to 12 hours
Drug concentration in plasma at 12 hours after administration (C12h) for tipranavir/ritonavir | up to 12 hours

SECONDARY OUTCOMES:
Maximum plasma concentration at steady state (Cmax,ss) | up to 24 hours
Trough plasma concentration at steady state (Cmin) | up to 24 hours
Mean residency time (MRT) | up to 24 hours
Apparent terminal half life (T1/2) | up to 24 hours
Time of maximum concentration (Tmax) | up to 24 hours
Oral clearance (CL/F) | up to 24 hours
Apparent volume of distribution during the terminal elimination phase, divided by F (bioavailability factor) (Vz/F) | up to 24 hours
Number of subjects with clinically significant findings in vital signs (pulse rate, blood pressure) | up to 14 days
Number of subjects with clinically significant findings in physical examination | up to 14 days
Number of subjects with clinically significant findings in electrocardiogram | up to 14 days
Number of subjects with clinically significant findings in laboratory tests | up to 14 days
Number of subjects with adverse events | up to 14 days